CLINICAL TRIAL: NCT01467284
Title: School Worksite Weight Gain Prevention Intervention Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Stephenie Lemon, Associate Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01CA132941 (NIH)
Record Dates: First submitted 2011-10-07; First posted 2011-11-08 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Obesity
Keywords: Obesity; Workplace; Intervention; Diet; Exercise
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Step Ahead (Experimental): Promotion of weight gain prevention among teachers and staff in public high schools through Step Ahead, a comprehensive intervention targeting three levels suggested by the ecological framework health behavior change: organizational school level, interpersonal level, and individual level.
  Interventions: Behavioral: Step Ahead
- Basic Intervention (Active Comparator): Promotion of weight gain prevention among teachers and staff in public high schools through receipt of the workbook print materials and access to website similar to the enhanced intervention.
  Interventions: Behavioral: Basic Intervention

INTERVENTIONS:
Behavioral: Step Ahead — Promotion of weight gain prevention among teachers and staff in public high schools through Step Ahead, a comprehensive intervention targeting three levels suggested by the ecological framework health behavior change: organizational school level, interpersonal level, and individual level.
  Arms: Step Ahead
Behavioral: Basic Intervention — Promotion of weight gain prevention among teachers and staff in public high schools through receipt of the workbook print materials and access to website similar to the enhanced intervention.
  Arms: Basic Intervention

SUMMARY:
The proposed site-level randomized trial will test the effectiveness of a work site intervention based on an ecological framework at preventing weight gain among high school employees in Massachusetts. The investigators hypothesis is that the intervention will positively impact healthy dietary patterns and physical activity, perceived organizational commitment, coworker influences, social support, self-efficacy, and self-control, which in turn will positively mediate or moderate the positive associations between the intervention and the primary outcomes (change in weight, BMI, and waist circumference). If effective, the intervention is designed to be generalizable to high school settings across the country and has the potential to reduce the morbidity, mortality and economic costs of overweight and obesity in this important population.

ELIGIBILITY:
Inclusion Criteria:

* work at least 15 hours per week, or approximately half of the school week,
* only work at one school participating in the study,
* not be in a "leadership" position in the school (e.g. principals and vice-principals)
* be able to stand up
* speak English
* plan to be employed at the school for the next 24 months

Exclusion Criteria:

* work less than 15 hours per week
* work at more than one participating school
* work in a "leadership" position (e.g. principal or vice-principal)
* does not speak English
* unable to stand up

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 844 (Actual)
Dates: Start 2009-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
High school employee change in weight | 24 months post-baseline
  Test the effectiveness of a worksite intervention based on an ecological framework at preventing an increase in weight among high school employees in Massachusetts

SECONDARY OUTCOMES:
High school employee change in BMI | 24 months post-baseline
  Test the effectiveness of a worksite intervention based on an ecological framework at preventing an increase in BMI among high school employees in Massachusetts
High School employee change in waist circumference | 23 months post-baseline
  Test the effectiveness of a worksite intervention based on an ecological framework at preventing an increase in waist circumference among high school employees in Massachusetts
Weight management behaviors | 24 months post-baseline
  Test the effectiveness of a worksite intervention compared to the control condition on physical activity and healthy eating behaviors among high school employees in Massachusetts.
High school employee absenteeism | 24 months post-baseline
  Test the effectiveness of a work site intervention based on an ecological framework at preventing absenteeism among high school employees in Massachusetts.

CONTACTS AND LOCATIONS:
Overall Officials: Stephenie Lemon, PhD, Principal Investigator — University of Massachusetts, Worcester; Lori Pbert, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

REFERENCES:
- [Derived] Wang ML, Haughton CF, Frisard C, Pbert L, Geer C, Lemon SC. Perceived weight status and weight change among a U.S. adult sample. Obesity (Silver Spring). 2017 Jan;25(1):223-228. doi: 10.1002/oby.21685. Epub 2016 Nov 15. PMID 27863126
- [Derived] Alker HJ, Wang ML, Pbert L, Thorsen N, Lemon SC. Impact of school staff health on work productivity in secondary schools in Massachusetts. J Sch Health. 2015 Jun;85(6):398-404. doi: 10.1111/josh.12266. PMID 25877437